CLINICAL TRIAL: NCT02834481
Title: ANI/NIPE Assessment of Pain Monitoring With ANI (Analgesia Nociceptive Index)/NIPE (Newborn Infant Parasympathetic Evaluation) Monitor Program in Pediatric Cardiac Surgery Postoperative.
Brief Title: Assessment of Pain Monitoring With ANI/NIPE Monitor Program in Pediatric Cardiac Surgery Postoperative.
Acronym: ANI/NIPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: too complicated recruitment
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/15/7852
Record Dates: First submitted 2016-07-12; First posted 2016-07-15 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Pain
Keywords: Pain Care; Pediatric and Neonatal Intensive Care Units
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- : ventilated children (Other): ventilated children admitted in PICU postoperative of cardiac surgery with extracorporeal circulation with ANI/NIPE
  Interventions: Device: ANI/NIPE

INTERVENTIONS:
Device: ANI/NIPE — ANI/NIPE monitors is a continuous noninvasive measurement of the parasympathetic tone, as a component of the autonomous nervous system. It uses the tiny variations of heart rate induced by each respiratory cycle (natural or induced) to quantify parasympathetic tone (respiratory sinus arrhythmia).

SUMMARY:
The main objective is to assess correlation between ANI/NIPE values and external evaluation COMFORT B scale during painful medical cares and during said comfort medical cares in intubated children admitted in pediatric intensive care unit postoperative of cardiac surgery with extracorporeal circulation.

DETAILED DESCRIPTION:
ANI/NIPE monitors is a continuous noninvasive measurement of the parasympathetic tone, as a component of the autonomous nervous system. It uses the tiny variations of heart rate induced by each respiratory cycle (natural or induced) to quantify parasympathetic tone (respiratory sinus arrhythmia).

Developed in surgical units, the ANI monitor has rarely been studied in pediatrics (only 2 publications, and only concerning peroperative measures). The NIPE monitor has only been available since 2014. Nevertheless, adult surveys and fundamental scientific publications on heart rate variations suggest that these monitors can evaluate pain on a continuous way. No study has been led in pediatric intensive care units.

In our study, a continuous blinded monitoring will be set up as soon as patients' admittance for all eligible subjects. We will study, for children in cardiac post-surgery, ANI/ NIPE values and COMFORT B values during both painful and non-painful cares to determine correlation between those values. We will analyze a posteriori the ANI/NIPE values, through a standardized protocol, to recount the sequence of care and to determine discrepancies in drug consumption. Data gathering will be made in the first 48h after admittance in Pediatric Intensive Care Units (PICU). Patients will not be followed after leaving PICU.

ELIGIBILITY:
Inclusion Criteria:

* ventilated children admitted in PICU postoperative of cardiac surgery with extracorporeal circulation, consent of the parental control, children benefiting from social security system

Exclusion Criteria:

* Heart rhythm disorder, use of heart rhythm disorder treatments, use of active pacemaker, which make ANI/NIPE values impossible to interpret

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Comparison between ANI/NIPE values and COMFORT B scale values assessed by coefficient of correlation in patients upper than two years old and in patients under two years old | Through the study completion (24 months)
  coefficient correlation is used with confident interval of 95 per cent

SECONDARY OUTCOMES:
Determination of pain detection threshold with ANI/NIPE scale using receiving operator characteristics receiving operator characteristics (ROC) curve. | Through the study completion (24 months)
  In comparison with COMFORT B scale
Determination of pain detection threshold with COMFORT B scale using ROC curve. | Through the study completion (24 months)
  In comparison with ANI/NIPE scale
Evolution of ANI/NIPE value during pain care | Through the study completion (24 months)
  assessed by scale value
Evolution of ANI/NIPE value during comfort care | Through the study completion (24 months)
  assessed by scale value

CONTACTS AND LOCATIONS:
Overall Officials: PELLUAU Sonia, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No